CLINICAL TRIAL: NCT01339702
Title: Impact of Implementing the EMS Traumatic Brain Injury Treatment Guidelines
Brief Title: The EPIC Project: Impact of Implementing the EMS Traumatic Brain Injury Treatment Guidelines
Acronym: EPIC
Status: Completed | Type: Observational
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Daniel Spaite, Professor of Emergency Medicine, University of Arizona
Other Study IDs: EPIC-NINDS-R01NS071049
Record Dates: First submitted 2011-04-15; First posted 2011-04-21 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Brain Injuries, Traumatic; Injuries, Acute Brain; TBI (Traumatic Brain Injury)
Keywords: Traumatic Brain Injury; TBI; Head Trauma; Acute Traumatic Brain Injury; Trauma, Brain
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries; Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pre-implementation cohort ("before"): This cohort is a combination of retrospective and some prospective severe TBI patients cared for in the EMS systems of Arizona BEFORE implementation of the national prehospital TBI management guidelines
- Post-implementation cohort ("after"): This cohort is a comprised of prospective severe TBI patients cared for in the EMS systems of Arizona AFTER training EMS providers in the implementation of the national prehospital TBI management guidelines. It is intended that these patients will receive the "bundle" of care specified in the TBI Guidelines.
  Interventions: Other: The National Prehospital TBI Management Guidelines

INTERVENTIONS:
Other: The National Prehospital TBI Management Guidelines — In the post-implementation (after) cohort, implementation of the entire "bundle" of the TBI treatment guidelines with special emphasis on prevention and treatment of hypotension (IV crystalloids), prevention and treatment of hypoxia (pre-oxygenation with high-flow O2 via non-rebreather mask, bag-valve-mask, extraglottic airways/intubation when basic maneuvers have failed), and prevention of hyperventilation (in intubated patients) and prevention/treatment of hypoventilation (in all patients).
  Other Names: Brain Trauma Foundation TBI Guidelines; National Association of EMS Physicians TBI Guidelines
  Groups: Post-implementation cohort ("after")

SUMMARY:
Evaluation of the impact (on survival and other outcomes) of implementing the Brain Trauma Foundation/National Association of EMS Physicians Traumatic Brain Injury (TBI) guidelines in the prehospital EMS systems throughout the state of Arizona.

DETAILED DESCRIPTION:
* Significance: Approximately 1.4 million victims of Traumatic Brain Injury (TBI) are seen in emergency departments each year in the U.S. and, of those, 50,000 die and 235,000 are hospitalized. A least 2% of the U.S. population has a TBI-related long-term need for help to perform activities of daily living. There is growing evidence that the management of TBI in the early minutes after injury profoundly impacts outcome. This has led to the promulgation of evidence-based TBI treatment guidelines by authoritative national and international scientific bodies. Reports on guideline implementation in the hospital setting are very promising. However, no studies have evaluated their impact in the prehospital setting. While randomized prehospital trials to identify the effectiveness of the guidelines would clearly be optimal, the strong indirect evidence currently precludes withholding guideline therapy because of ethical considerations. Thus a large, prospective, historically controlled, observational study is the best methodology currently available to evaluate the effectiveness of implementing the guidelines in the prehospital setting.
* Specific Aim: To test the hypothesis that implementation of the TBI guidelines in a statewide EMS system will reduce mortality and improve non-mortality outcomes in adults and children with moderate to severe TBI.
* Objective #1: Implement the nationally-vetted TBI guidelines across a broad variety of EMS systems (urban, suburban and rural) throughout the State of Arizona. This will be accomplished through the statewide collaboration between the University of Arizona, the Arizona Department of Health Services, and local EMS agencies responding to 85% of the state's population. This will mirror the approach that has been successfully employed to study and document a tripling of patient survival from out-of-hospital cardiac arrest in the state.
* Objective #2: Collect prehospital EMS and trauma center data on severe TBI patients cared for by participating EMS agencies to determine pre-implementation and post-implementation injury severity/risk-adjustment measures and outcomes.
* Objective #3: Evaluate the impact of prehospital guideline implementation on the following outcomes: 1) Overall mortality (primary outcome), 2) mortality among patients who are intubated prior to hospital arrival, and 3) non-mortality outcomes such as hospital/intensive care unit length of stay, ventilator days, and patient disposition.
* Relevance/health impact: The societal burden of TBI is immense. While the potential for dramatically reducing morbidity and mortality by early treatment appears to be great, the effectiveness of the prehospital guidelines remains unproven. Demonstrating the impact of guideline therapy would potentially lead to widespread implementation of the effective interventions. This could dramatically reduce morbidity and mortality from this major public health problem. On the other hand, if the guidelines are not effective despite confirmed implementation across a wide variety of EMS systems throughout the entire state, this would provide the ethical basis for conducting future randomized trials.

ELIGIBILITY:
Inclusion Criteria:

* Adults and children with physical trauma who: 1) are transported directly to or are transferred to a level I TC by participating EMS agencies, 2) have hospital diagnosis(es) consistent with TBI (either isolated or multisystem trauma that includes TBI), and 3) meet at least one of the following definitions for severe TBI: a) last prehospital GCS or first hospital/trauma center GCS <9; b) AIS-head of ≥3, c) CDC Barell Matrix-Type 1, d) undergo prehospital ETI, nasal intubation, or cricothyrotomy.

Exclusion Criteria:

* Patients with brain injury from: 1) non-mechanical mechanisms (e.g., drowning); 2) choking, primary asphyxiation, or strangulation; 3) environmental injury (e.g., hyperthermia); 4) poisoning (e.g., drug overdose, carbon monoxide, insecticides); 5) intracranial hemorrhage of non-traumatic origin; 6) other non-traumatic, acute neurological emergencies (e.g., bacterial meningitis).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children of all ages with acute, moderate or severe TBI cared for in the participating EMS systems of Arizona who are taken to a Level 1 Trauma Center (either directly by EMS or transfered by EMS). This will include approximately 4 years of retrospective cases and 4.5 years of prospective cases.
Sampling Method: Probability Sample
Enrollment: 26873 (Actual)
Dates: Start 2011-09; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Survival | hospital discharge
  Participants will be followed for the duration of hospital stay. The average time from admission to either discharge or death is expected to be approximately 3 weeks.

SECONDARY OUTCOMES:
hospital length of stay | discharge from hospital
  This parameter will be the number of days that the patients spend in their initial, acute hospitalization. An average of 3 weeks is expected.
Intensive care unit length of stay | admission to ICU to transfer from ICU
  This parameter will be the number of days that the patients spend in the ICU. An average of 1 week is expected.
ventilator days | during hospitalization
  When applicable, the number of days a patient is on a ventilator. This is expected to be an average of 2 days among all patients and 1 week among the subgroup of patients who are placed on a ventilator.
Patient disposition | hospital discharge
  where the patient was discharged or transferred to (e.g., skilled nursing facility, home, rehabilitation hospital) (average 3 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W Spaite, MD, Principal Investigator — University of Arizona
Locations (1):
- Arizona Emergency Medicine Research Center, Phoenix, Arizona, United States

REFERENCES:
- [Background] Spaite DW, Bobrow BJ, Stolz U, Sherrill D, Chikani V, Barnhart B, Sotelo M, Gaither JB, Viscusi C, Adelson PD, Denninghoff KR. Evaluation of the impact of implementing the emergency medical services traumatic brain injury guidelines in Arizona: the Excellence in Prehospital Injury Care (EPIC) study methodology. Acad Emerg Med. 2014 Jul;21(7):818-30. doi: 10.1111/acem.12411. Epub 2014 Aug 11. PMID 25112451
- [Derived] Spaite DW, Hu C, Bobrow BJ, Barnhart B, Chikani V, Gaither JB, Denninghoff KR, Bradley GH, Rice AD, Howard JT, Keim SM. Optimal Out-of-Hospital Blood Pressure in Major Traumatic Brain Injury: A Challenge to the Current Understanding of Hypotension. Ann Emerg Med. 2022 Jul;80(1):46-59. doi: 10.1016/j.annemergmed.2022.01.045. Epub 2022 Mar 24. PMID 35339285
- [Derived] Gaither JB, Spaite DW, Bobrow BJ, Keim SM, Barnhart BJ, Chikani V, Sherrill D, Denninghoff KR, Mullins T, Adelson PD, Rice AD, Viscusi C, Hu C. Effect of Implementing the Out-of-Hospital Traumatic Brain Injury Treatment Guidelines: The Excellence in Prehospital Injury Care for Children Study (EPIC4Kids). Ann Emerg Med. 2021 Feb;77(2):139-153. doi: 10.1016/j.annemergmed.2020.09.435. Epub 2020 Nov 11. PMID 33187749
- [Derived] Spaite DW, Bobrow BJ, Keim SM, Barnhart B, Chikani V, Gaither JB, Sherrill D, Denninghoff KR, Mullins T, Adelson PD, Rice AD, Viscusi C, Hu C. Association of Statewide Implementation of the Prehospital Traumatic Brain Injury Treatment Guidelines With Patient Survival Following Traumatic Brain Injury: The Excellence in Prehospital Injury Care (EPIC) Study. JAMA Surg. 2019 Jul 1;154(7):e191152. doi: 10.1001/jamasurg.2019.1152. Epub 2019 Jul 17. PMID 31066879
- [Derived] Spaite DW, Hu C, Bobrow BJ, Chikani V, Barnhart B, Gaither JB, Denninghoff KR, Adelson PD, Keim SM, Viscusi C, Mullins T, Sherrill D. The Effect of Combined Out-of-Hospital Hypotension and Hypoxia on Mortality in Major Traumatic Brain Injury. Ann Emerg Med. 2017 Jan;69(1):62-72. doi: 10.1016/j.annemergmed.2016.08.007. Epub 2016 Sep 28. PMID 27692683